CLINICAL TRIAL: NCT01401855
Title: Optical Probe In Thyroid Cancer
Brief Title: Use of an In Vivo Optical Probe to Discriminate Benign From Malignant Thyroid Nodules
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: Fraunhofer USA (Unknown)
Responsible Party: Principal Investigator, Stephanie Lee, Assistant Professor of Medicine, Boston Medical Center
Other Study IDs: H-29527
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Cancer; Thyroid
Keywords: Diagnosis; Fine Needle Aspiration Biopsy
MeSH Terms: conditions — Neoplasms; Thyroid Diseases; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- In Vivo Probe Prediction
- Cytology Results

SUMMARY:
This study will investigate the usefulness of an optical probe in the differentiation of thyroid cancer from normal thyroid tissue in a thyroidectomy specimen. This is the next step in the research that this team has conducted through our prior Institutional Review Board (IRB)H-28135, in which the investigators successfully demonstrated that use of the optical probe readings on thyroid specimens ex vivo could successfully discriminate benign from malignant disease. The Elastic Scattering Spectroscopy (ESS) probe has also been IRB approved and a clinical trial conducted in vivo at Boston University/Boston Medical Center by Dr. Satish Singh and Dr. Irving Bigio. The investigators intend to now bring this project to the clinical setting of thyroid disease. The optical real-time readings will be compared to the histological analysis from the same area. Subjects already undergoing thyroid biopsy for thyroid disease including thyroid nodules, thyroid cancer and thyroid goiter with nodules will be eligible to participate. During the already scheduled thyroid procedure using a fine needle aspiration biopsy needle, optical readings will be taken from the thyroid gland and these same areas will then be analyzed in the usual standard fashion. The reading will then be correlated with the histological results. In addition, if lymph nodes are biopsied as part of the evaluation they will also be tested prior to histological standard processing. All specimens and data will be de-identified once data collection and analysis is complete. Our goal is to use optical real-time readings to improve the differential diagnosis of benign from malignant thyroid nodules and avoid surgery for the purpose of diagnosis alone.

DETAILED DESCRIPTION:
Background: Thyroid cancer is the most common endocrine malignancy. The current gold standard, fine-needle aspiration (FNA) biopsy, yields approximately 10-25% of indeterminate results, leading to patients undergoing thyroidectomy for diagnosis. Elastic scattering spectroscopy (ESS) is a new, minimally invasive optical-biopsy technique, mediated by fiber-optic probes, that which is sensitive to cellular and sub-cellular morphological features. We assessed the potential to incorporate an ESS probe into a 23-gauge needle biopsy to use in preoperative trans-cutaneous biopsy of the thyroid to differentiate benign from malignant thyroid nodules.

Methods: We designed and built a miniaturized ESS probe that can fit through a 23-gauge biopsy needle and tested it under an IRB-approved protocol on 34 patients undergoing ultrasound-guided FNA biopsy of thyroid nodules in the endocrine clinic. ESS data was collected during the conduct of their biopsy using optical 5 repetitive readings from three distinct locations within the thyroid nodule. Using cytology as our gold standard, spectral analyses were compared between benign and malignant thyroid nodules. For indeterminate cytology, final post-surgery pathology of the tissue was used for the comparison.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing thyroid biopsy for thyroid nodules, thyroid cancer, and thyroid goiter with nodules. Only those patients requiring sampling under established standard of care criteria and already scheduled to undergo biopsy for clinical purposes will undergo optical biopsy at the same time as their physical biopsy.

Exclusion Criteria:

* Subjects with nodules smaller than 1 cm, infectious diseases, on medication (such as coumadin) that may interfere with optical readings

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects, male and female, undergoing thyroid fine needle aspiration biopsy at Boston Medical Center ages 18 and older. Study population includes all ethnic groups.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Assess optical probe for the differentiation of thyroid cancer from normal thyroid tissue and benign thyroid nodules | 2 years
  The objective is to assess a device called an optical probe for the differentiation of thyroid cancer from normal thyroid tissue, benign thyroid nodules or parathyroid glands, and the detection of thyroid cancer within lymph nodes. The gold standard for diagnosis is ultrasound guided fine needle aspiration biopsy of the nodule. Based on cytology from Fine Needle Aspiration (FNA), 10% of nodules are cancer, 70% are benign (not cancer) and 20% are "indeterminate." The proposed device aims to decrease the number of patients that undergo surgery for diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rosen, MD/FACS, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States